CLINICAL TRIAL: NCT04711928
Title: Do Trained Athletes Also Suffer From the Sedentary Behaviour Paradigm?: the Association Between Sedentary Behaviour and Cardiometabolic Health
Brief Title: The Association Between Sedentary Behaviour and Cardiometabolic Health in Trained Athletes
Acronym: HPAC
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Bert Op't Eijnde, Professor, Hasselt University
Other Study IDs: CME2020/012
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Cardiometabolic Health; Sedentary Behavior; Physical Activity; Athletes
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trained athletes: Active individuals with at least 4 training hours per week.
  Interventions: Behavioral: Physical activity and sedentary behaviour

INTERVENTIONS:
Behavioral: Physical activity and sedentary behaviour — Athletes with a high physical activity and a low or high sedentary time

SUMMARY:
Physical inactivity is one of the major contributing factors for the development of chronic diseases and highly correlated with increased all-cause mortality. In the last decade an exponential growth in research concerned with the study of sedentary behaviour and the potential for detrimental effects on health have been published. In this field increasing evidence suggests that prolonged periods of sedentary time, independent of the amount of physical activity, also increases the risk for the development of several chronic conditions and all-cause mortality. Here, sedentary behaviour is defined as "any waking behaviour, characterized by a low energy expenditure (≤1.5 METs), while being in a sitting or reclining posture". Interestingly, the advised moderate-to-vigorous bouts of exercise recommended by the various guidelines cannot compensate the negative impact on health risks arising from prolonged periods of sitting. In other words, it seems that people compensate their total amount of physical activity after exercise training by decreasing their physical activity levels throughout the rest of the day. Here, it appears that frequent, even low-intensity interruptions of periods of sitting are required for good cardiometabolic health. Therefore, not only physical activity but also prolonged sitting should be targeted to optimize cardiometabolic health. Nevertheless, a recent harmonized meta-syntheses indicated that the association between self-reported sitting with all-cause and cardiovascular disease mortality are only partially independent of physical activity, but were particularly evident in those who undertake insufficient physical activity (<150min/week). However, it is unclear whether high amounts of objectively measured physical activity attenuates or even eliminates the detrimental effects of prolonged sitting. In addition, it is still unclear whether high amounts of physical activity can preserve a healthy cardiometabolic risk profile, despite prolonged sitting. Therefore, in this study we want to investigate the association between sedentary behaviour, physical activity and cardiometabolic health in highly physically active adults.

ELIGIBILITY:
Inclusion Criteria:

* Active individuals with at least 4 training hours per week

Exclusion Criteria:

* pregnancy
* Any known contradiction for physical activity
* Systolic blood pressure >160mmHg, diastolic blood pressure >100mmHg
* More than 20 alcohol consumptions per week
* Participants diagnosed with any known chronic disease

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Active individuals with at least 4 training hours per week and between 18 and 45 years of age.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Sedentary time (min/day) | day 1
  Main outcome parameter of sedentary behaviour indication measured with ActivPAL3

SECONDARY OUTCOMES:
Moderate-to-vigorous physical activity time (min/day) | day 1
  Physical activity parameter measured with ActivPAL3
Light physical activity time (min/day) | day 1
  Physical activity parameter measured with ActivPAL3
Blood glucose concentration | day 1
  Parameter of glucose homeostatis
Blood insulin concentration | day1
  Parameter of glucose homeostatis
Blood total cholesterol concentration | day 1
  Parameter of lipid metabolism
Blood triglyceride concentration | day 1
  Parameter of lipid metabolism
Blood high density lipoprotein concentration | day 1
  Parameter of lipid metabolism
Blood low density lipoprotein concentration | day 1
  Parameter of lipid metabolism
Fat mass (kg) | day 1
  Parameter of body composition measured with DEXA-scan
Lean mass (kg) | day 1
  Parameter of body composition measured with DEXA-scan
Systolic blood pressure | day 1
  Parameter of cardiovascular health
Diastolic blood pressure | day 1
  Parameter of cardiovascular health
Maximal oxygen uptake | day 1
  Parameter of oxygen capacity measured with cardiopulmonary exercise testing

CONTACTS AND LOCATIONS:
Locations (1):
- Wouter Franssen, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franssen WMA, Jermei J, Savelberg HHCM, Eijnde BO. The potential harms of sedentary behaviour on cardiometabolic health are mitigated in highly active adults: a compositional data analysis. J Act Sedentary Sleep Behav. 2023 Mar 2;2(1):6. doi: 10.1186/s44167-023-00015-7. PMID 40217441